CLINICAL TRIAL: NCT04971460
Title: The Mental Well-being of Fathers and Partners of Women Accessing Perinatal Mental Health Services
Brief Title: The Mental Well-being of Fathers and Partners
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 291920
Record Dates: First submitted 2021-05-10; First posted 2021-07-21 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2021-04

CONDITIONS: Mental Health Disorder; Fathers
Keywords: Fathers; Perinatal
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mother and Baby Unit: Fathers and partners of women admitted to a Mother and Baby Unit
- Peri-natal Community Mental Health Services: Fathers and partners of women accessing community perinatal mental health services
- Control group: Fathers and partners of women who are not accessing mental health services in the perinatal period

SUMMARY:
The purpose of this study is to assess the acceptability and feasibility of screening common mental health difficulties in fathers and partners of women accessing perinatal mental health services.

DETAILED DESCRIPTION:
Where women have mental health disorders, this can put significant strain on their partners. As well as supporting the mother and dealing with worries and uncertainty about her wellbeing, partners may take on additional childcare and household duties alongside maintaining work commitments. As a result, mental health professionals are considering ways to involve and support partners and other family members where women are accessing specialist services.

This feasibility study will involve the screening of fathers/partners of women accessing perinatal mental health services, for mental health disorders including depression, anxiety disorders and post-traumatic stress disorder (PTSD). Previous empirical evidence has largely focussed on fathers but we will include partners i.e., whoever the mother identifies as her partner, therefore including individuals in same sex relationships or when the main partner is a stepparent. The screening questionnaires will help us to understand the mental health needs of fathers/partners of women who are being cared for by perinatal mental health services. This will also help us see if partners find it acceptable to complete questionnaires on their mental health and family functioning online.

Three groups of participants will be approached across a 6-month period. The first; fathers/partners of women being treated in a Mother and Baby Unit. The second; fathers/partners of women being treated in community services (i.e. community Perinatal Mental Health Services). The third; fathers/partners of women who have not experienced mental health difficulties in the perinatal period.

Fathers/partners in the clinical groups will initially be approached by clinicians in the relevant service (Mother and Baby Unit or Community Perinatal Mental Health Teams). They will be asked for verbal consent to be contacted by the research team. The research team will then contact the participant and provide further information about the study and obtain informed consent. Participants in the control group will be recruited online via social media and through local charities and community groups.

Fathers/partners will be invited to complete screening questionnaires on their mental wellbeing -(the Edinburgh Post-natal Depression Scale (EPDS), the Gotland Male Depression Scale, the Generalised Anxiety Disorder-7 scale (GAD-7), the City Birth Trauma Scale), a demographic questionnaire and the Couple's Satisfaction Index. Participants will be able to complete these questionnaires online or via hard copies.

The study will help to inform our understanding of whether fathers/partners find it acceptable to complete mental health screening questionnaires. It will also help to identify if fathers/partners are more at risk of developing mental health difficulties if the mother is also experiencing a mental health difficulty.

ELIGIBILITY:
Inclusion Criteria:

Fathers and partners of women:

1. Admitted to the SLaM Mother and Baby Unit or
2. Seen by SLaM Community Perinatal Mental Health services or
3. Not accessing a mental health service currently or during the perinatal period (pregnancy to 12-months postpartum).

   * Biological father, step-father, same sex partner or any other adult that identifies as the woman's 'primary' partner.
   * Women who are pregnant or up to 12-months post-partum
   * Adult fathers/partner aged 18 years and above
   * Father/partner has proficient level of English to complete screening questionnaires.
   * Father/partner has the ability to complete questionnaires electronically on a phone/table/computer or to complete paper questionnaires
   * Father/partner is able to give informed consent and comply with study procedures

Exclusion Criteria:

Fathers and partners

* Unable to provide consent to complete questionnaires Women
* In the 'healthy' group - if the mother is accessing mental health services or has done during the perinatal period (pregnancy to 12-months postpartum) Infant offspring
* Aged over 12 months

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Three groups of fathers/partners will be invited to take part in the study - fathers/partners of women being treated in a mother and baby unit, fathers/partners of women being treated in community services and fathers/partners of women who are not accessing mental health services. Participants will be recruited via the SLaM Mother and Baby Unit and Community perinatal teams. The community sample will be recruited online via social media and through local community groups/charities. Fathers/partners in the community sample will be asked to confirm that the mother is not currently accessing mental health services and hasn't accessed mental health services during the perinatal period (pregnancy to 12-months post-partum).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-07-24 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
How many partners/fathers complete the screening questionnaires | 6-months
  How many partners/fathers complete the screening questionnaires online over the 6-month recruitment period.

SECONDARY OUTCOMES:
Prevalence of mental health difficulties | 6-months
  To estimate the prevalence of common mental health difficulties in three study groups:
  1. fathers and partners of women admitted to a Mother and Baby Unit
  2. fathers and partners of women accessing community perinatal mental health services
  3. fathers and partners of women who are not accessing mental health services in the perinatal period

CONTACTS AND LOCATIONS:
Overall Officials: Vaheshta Sethna, DPhil, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No